# **Informed Consent Form**

Title: Smoke-free Air Coalitions in Georgia and Armenia: A Community

**Randomized Trial** 

NCT Number: NCT03447912

**IRB Approval Date:** November 11, 2022

# Emory University Consent To Enroll in Research Study

Title: Smoke-free Air Coalitions in Georgia and Armenia: A Community Randomized Trial

<u>Principal Investigator:</u> This study is being conducted by Carla Berg, PhD, Michelle Kegler, PhD, Department of Behavioral Sciences and Health Education, Rollins School of Public Health, Emory University.

Funding Source: Pending funding from the US National Institutes of Health Fogarty International Center.

### Introduction

You are being asked to be in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. You can skip any questions that you do not wish to answer.

Before making your decision:

- Please carefully read this form or have it read to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. By signing this form you will not give up any legal rights.

#### **Study Overview**

The purpose of this study is to examine factors related to tobacco use in your community as well as your own experiences with tobacco.

# **Procedures**

If you agree, you will complete a 15-20 minute, one-time written survey in either English or your native language of [insert language]. We anticipate that roughly 50 individuals per community will participate in this study, and 28 communities overall will participate (total 1,400 participants overall).

# **Risks and Discomforts**

The major risk of this study is loss of privacy and confidentiality of the information. However, participants will be assigned a study ID number, assuring that no personal identifying information will be linked directly with the data. A separate key linking participant ID to personal identifying information will be encrypted and stored.

## **Benefits**

There are no anticipated benefits to participation, but we may learn valuable information that can be used to improve the health of others.

# Compensation

There is no compensation for participating in this study.

#### Confidentiality

Certain offices and people other than the researchers may look at study records. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include [the Office for

Page 1 of 3 IRB Form 05022016 Version Date: 05/02/2016

Document Approved On: 4/23/2019

IRB00097093 IRB Approved

# **Emory University IRB** IRB use only

Study No.: IRB00097093 Document Approved On: 4/23/2019

Human Research Protections, the funder(s), the Emory Institutional Review Board, the Emory Office of Research Compliance]. Study funders may also look at your study records. Emory will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

Study records can be opened by court order. They may also be produced in response to a subpoena or a request for production of documents.

# **Voluntary Participation and Withdrawal from the Study**

You have the right to leave a study at any time without penalty. You may refuse to do any procedures you do not feel comfortable with, or answer any questions that you do not wish to answer.

The researchers and funder also have the right to stop your participation in this study without your consent if they believe it is in your best interest

# **Contact Information**

Contact Carla Berg at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at 404-712-0720 or irb@emory.edu:

- if you have questions about your rights as a research participant.
- if you have guestions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at http://www.surveymonkey.com/s/6ZDMW75.

Version Date: 05/02/2016

IRB00097093 IRB Approved 11/11/2022 Study No.: IRB00097093

Signature of Subject

Signature of Person Conducting Informed Consent Discussion

# Emory University IRB IRB use only

Consent
Please, print your name and sign below if you agree to be in this study. By signing this consent form, you will not give up any of your legal rights. We will give you a copy of the signed consent, to keep.

Name of Subject

Document Approved On: 4/23/2019

Date

Date

Time

Time

Page 3 of 3 Version Date: 05/02/2016